CLINICAL TRIAL: NCT06612905
Title: Effect Of Social Media On Body Weight And Eating Behaviour In Housewife Versus Worker Postmenopausal Women
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Reda Mahmoud, Principal Investigator, Cairo University
Other Study IDs: P.T.REC/012/004515
Record Dates: First submitted 2024-09-22; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Social Media Addiction
MeSH Terms: conditions — Internet Addiction Disorder | interventions — Basal Metabolism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Housewife postmenopausal women: It will consist of 74 housewife postmenopausal women, at least 12 months after their last menstrual cycle.
  Interventions: Other: Detection of the time spent on social media; Other: Evaluation of body composition and basal metabolic rate; Other: Evaluation of eating behavior among social media users
- Worker postmenopausal women: It will consist of 74 worker postmenopausal women, at least 12 months after their last menstrual cycle.
  Interventions: Other: Detection of the time spent on social media; Other: Evaluation of body composition and basal metabolic rate; Other: Evaluation of eating behavior among social media users

INTERVENTIONS:
Other: Detection of the time spent on social media — The time spent on social media will be assessed by using the social networking usage questionnaire (SONTUS) for all women in both groups (A and B).
Other: Evaluation of body composition and basal metabolic rate — They will be evaluated using Inbody (Bodecoder)(CHL-818, made in China) and its software (2.2.1 apk)
Other: Evaluation of eating behavior among social media users — Scale of effects of social media on eating behavior (SESMEB) will be used for all women in both groups (A and B) to assess the effect of social media on their eating behavior. The SESMEB consists of one subscale and eighteen items. It is a reliable and valid scale, items scale is evaluated with five-point Likert scale. Each item is evaluated as 'always' five points, 'often' four points, 'sometimes' three points, 'seldom' two points and 'never' one point. There is no reverse coded substance. As it is mentioned in item analysis part, total score can be calculated. According to this minimum eighteen and maximum ninety points from SESMEB scale can be taken as total point. As a result, the increase in the person's scale score means that the level of being affected by the eating media increases.

SUMMARY:
The purpose of this study is to determine the effect of social media on body weight and eating behaviour in housewife versus worker postmenopausal women.

DETAILED DESCRIPTION:
Menopause altered fat distribution that occurs as negative impacts of the increase in insulin resistance, and the incidence of diabetes has risen exponentially. This increase, in turn, has been translates into an increased risk of cardiovascular disorder (CVD) and death, with the impact being greater in women than in men.

Media has been largely implicated in the widespread incidence of disordered eating worldwide. One of the main theories to explain the relationship between media and disordered eating is the sociocultural model. According to sociocultural theory, when young women are exposed to idealized body images in the media, they internalize these images gradually developing unrealistic body image expectations. In turn, failure to attain this idealized body image may result in body shape concerns, body dissatisfaction, and disordered eating behaviors.

Social media users are often exposed to advice and recommendations on diet and health issues through books, journals and electronic formats supported by a quick exchange of ideas through social media without scientific basis. The constant infiltration of social media into our life has necessitated a research on the effects of it on eating behavior. Owing to the prevalence of social media use, including the sharing photographs and making comments to foods, menus and recipes, it is especially important to identify the potential effects of these issues on eating behaviors.

People who use social media more are at greater risk of sleep disturbance that leads to obesity. It was reported that 40% decrease in weight gaining accrued in people who limits their screen-time than in people without such limitation.

There is widespread theoretical and practical interest in understanding how social media affect health related behaviours. Large observational studies of population health have discussed the effect of social media effect on human health even its benefits or hazards.

Previous studies illustrated the link between the time spent at social media and the resulted weight among young generations and adults, but to our knowledge, there is no previous study investigated the effect of social media on weight and eating behaviour among postmenopausal women or compared between workers and housewife postmenopausal women as regard to time spent on social media. So, this study will be the first one in this issue. Therefore, this study will be of valuable benefits and increased body knowledge of physical therapists in scientific field.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (housewifes/workers) at least 12 months of menstrual cessation will be included in this study.
* Their ages will range from 50 to 60 years old.
* They will be categorized as average to heavy users of social media according to (social networking usage questionnaire (SONTUS).
* The selected social media websites in this study will be Facebook, YouTube, what's app, Google chrome and Internet explorer.

Exclusion Criteria:

* Systematic disease (uncontrolled hypertension, diabetes mellitus).
* Thyroid, liver and kidney dysfunctions.
* Psycatric disorders
* Women received any hormonal therapy or received corticosteroids in the last six months prior the study

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: This study will be conducted on 148 post-menopausal women (workers/ housewives) at least one year after their last period. They will be selected from the outpatient clinic of women's health, Mataria Teaching Hospital, Cairo, Egypt.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-10 (Estimated)

PRIMARY OUTCOMES:
Detection of the time spent on social media | one month
  The time spent on social media will be assessed by using the social networking usage questionnaire (SONTUS) for all women in both groups (A and B). A complete and full demonstration for all items of the scale should be given to each women confirming on the importance of being honest in the scoring stage and all items should be scored as they will give us the true result. If any woman doesn't understand any item, they shouldn't give the item any score till they understand it. After finishing the scoring, the result will be interpreted, and according to it we will detect the type of social media user. In scoring the SONTUS, five component scores will be derived, then they will be summed to produce a global score that ranges from 5 to 23 and according the scores, the social media users will be classified as (low user, average user, high user, and extremely high user). An individual with a global score ranging from 5 to 9 is considered a low user of social networking sites (SNSs), while a
Measurement of body weight | one month
  It will be measured for all women in both groups, using Inbody (Bodecoder) (CHL-818, made in China) and its software (2.2.1 apk).
Calculation of body mass index (BMI) | one month
  It will be calculated for all women in both groups according to the following equation:
  BMI = (weight in kg)/(height in m^2 )
Measurement of total body fat | one month
  It will be measured for all women in both groups, using Inbody (Bodecoder) (CHL-818, made in China) and its software (2.2.1 apk).
Measurement of visceral fat | one month
  It will be measured for all women in both groups, using Inbody (Bodecoder) (CHL-818, made in China) and its software (2.2.1 apk).
Measurement of basal metabolic rate (BMR) | one month
  It will be measured for all women in both groups, using Inbody (Bodecoder) (CHL-818, made in China) and its software (2.2.1 apk).
Evaluation of eating behavior among social media users | one month
  Scale of effects of social media on eating behavior (SESMEB) will be used for all women in both groups to assess the effect of social media on their eating behavior. The SESMEB consists of one subscale and eighteen items. It is a reliable and valid scale, items scale is evaluated with five-point Likert scale. Each item is evaluated as 'always' five points, 'often' four points, 'sometimes' three points, 'seldom' two points and 'never' one point. There is no reverse coded substance. As it is mentioned in item analysis part, total score can be calculated. According to this minimum eighteen and maximum ninety points from SESMEB scale can be taken as total point. As a result, the increase in the person's scale score means that the level of being affected by the eating media increases.

CONTACTS AND LOCATIONS:
Overall Officials: Hala Mohamed Hanfy, PhD, Study Chair — Professor, Cairo university
Locations (1):
- Cairo University, Giza, Egypt